CLINICAL TRIAL: NCT00639327
Title: Randomized Phase II/III Trial of Second Line Chemotherapy Comparing CPT-11 Monotherapy Versus S-1/CPT-11 Combination for S-1 Refractory Gastric Cancer
Brief Title: Second Line Chemotherapy for S-1 Refractory Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Japan Clinical Cancer Research Organization (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Masashi Fujii/Associate Professor, Department of Digestive Surgery, Surugadai Nihon University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JACCRO GC-05
Record Dates: First submitted 2008-03-05; First posted 2008-03-20 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Gastric Cancer
Keywords: Stomach Neoplasms; Second line chemotherapy; Refractory to S-1; irinotecan; S-1 and Irinotecan Combination; Phase III study
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Irinotecan; titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): CPT-11+ S-1
  Interventions: Drug: S-1 + irinotecan
- B (Active Comparator): CPT-11
  Interventions: Drug: irinotecan

INTERVENTIONS:
Drug: S-1 + irinotecan — Irinotecan 150mg/m2 iv on day one and S-1 po days 1 to 14 every 3 weeks until PD
  Other Names: TS-1; CPT-11
  Arms: A
Drug: irinotecan — Irinotecan 150mg/m2 iv on day one every two weeks until PD
  Other Names: CPT-11
  Arms: B

SUMMARY:
The purpose of this study is compare overall survival of the test arm (CPT-11/S-1 combination) to the control arm (CPT-11 alone) in the subjects with S-1 refractory advanced gastric cancer.

DETAILED DESCRIPTION:
Standard chemotherapy for advanced gastric cancer (AGC) in the US is Cisplatin/5-FU (CF) or docetaxel/CF (DCF), is in Europe epirubicin/CF (ECF) or epirubicin/oxaliplatin/ capecitabine (EOX). Until 2006, there was no evidence of standard chemotherapy for AGC in Japan. In 2007, by the results of JCOG9912 trial (5-FU alone vs. CPT-11/CDDP vs S-1) and SPIRITS trial (S-1 alone vs. S-1/CDDP), S-1/CDDP is regarded as a new standard regimen in Japan. In 2008, by the results of TOP-002 trial (s-1 alone vs. S-1/CPT-11), S-1/CPT-11 could not show the superiority to S-1 alone. One of the other phase III trials, JACCRO GC-03 trial (S-1 alone vs. S-1/docetaxel, NCT00287768) is now ongoing. However, the position of CPT-11 in the treatment of AGC will be regarded as a second-line.

In Japan there is a controversy for the treatment of S-1 refractory gastric cancer. The controversy is continuing S-1 (like FOLFOX to FOLFIRI) or not as a second-line. After the successful adjuvant S-1 results (ACTS-GC trial), the same problem will occur in the patients who are recurrent from adjuvant S-1.

Then, we conducted a phase II/III trial of CPT-11 with or without S-1 in the treatment of first-line S-1 refractory AGC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven inoperable advanced gastric adenocarcinoma (including adenocarcinoma of the gastroesophageal junction) or relapse gastric adenocarcinoma
* Subjects must be able to take orally
* Subjects must be confirmed to be PD status by picture diagnosis after first-line chemotherapy using S-1 alone, S-1 + Cisplatinum or S-1 + taxane, except S-1 + CPT-11
* Within 4 weeks from the diagnosis of PD
* Total dosage of S-1 at the first-line is over 2,240mg/m2 in S-1 alone treatment, 1,680mg/m2 in the S-1 combination
* ECOG performance status ≤ 1
* Follow up Age 20 or over
* Life expectancy estimated more than 12 weeks
* Hgb ≥ 8 g/dL, WBC 4,000-12,000/mm3, ANC ≥ 2,000/mm3, platelets ≥ 100,000/mm3
* Creatinine ≤ upper normal limit (UNL)
* Total bilirubin ≤ 1.5 X UNL
* Written informed consent

Exclusion Criteria:

* S-1 + CPT-11 was employed as a first-line
* Any other cytotoxic agents therapy, immuno-therapy, radiation-therapy
* After S-1 adjuvant
* Suspended cases by adverse events by S-1 or S-1 combination
* Excessive amounts of ascites require drainage
* Known brain metastases
* History of hypersensitivity to fluoropyrimidines and CPT-11
* Pregnancy or lactation women, or women with suspected pregnancy or men with willing to get pregnant
* Active double cancer
* Gastrointestinal bleeding
* Any subject judged by the investigator to be unfit for any reason to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
In phase II part, progressive disease rate will be measured for the safety. In phase III part, overall survival will be measured for the benefit of doublet. | Phase II: 6 weeks from treatment, Phase III: 2 years OS from randomization

SECONDARY OUTCOMES:
Adverse events, response rates, progression free survival, time to treatment failure, change over rates to 3rd line | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Masashi Fujii, M.D.,PhD, Principal Investigator — Surugadai Nihon University Hospital
Locations (86):
- Japan (86):
  - Midori Municipal Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Aichi Medical University Hospital, Okazaki, Aichi-ken
  - Nakadoori General Hospital, Akita, Akita
  - Yamamoto Hospital, Noshiro, Akita
  - Aomori Prefectural Central Hospital, Aomori, Aomori
  - Hirosahi University Graduate School of Medicine, Hirosaki, Aomori
  - ChibaUniversity Hospital, Chiba, Chiba
  - Fukui Red Cross Hospital, Fukui-shi, Fukui
  - Saiseikai Hospital, Fukui-shi, Fukui
  - University of Fukui Faculty of Medical Scieneces Hospital, Yoshida-gun, Fukui
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - National Kyusyu Cancer Center, Fukuoka, Fukuoka
  - Kyusyu University Faculty of Medical Sciences, Fukuoka, Fukuoka
  - Nippon Steel Yawata Memorial Hospital, Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Fukushima Medical University, Fukushima, Fukushima
  - Gifu Municipal Hospital, Gifu, Gifu
  - Gifu Prefectural General Medical Center, Gifu, Gifu
  - Graduate School of Medicine, Gifu University, Gifu, Gifu
  - Gunma University Hospital, Maehashi, Gunma
  - Gunma Prefectural Cancer Center, Oota, Gunma
  - Fukuyama City Hospital, Fukuyama, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hiroshima University Research Institute for Radiation Biology and Medicine Tumor Surgery, Hiroshima, Hiroshima
  - Asahikawa Medical College Department Medicine, Asahikawa, Hokkaido
  - Asahikawa Medical College Hospital, Asahikawa, Hokkaido
  - Hakodate Goryoukaku Hopsital, Hakodate, Hokkaido
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hyogo Prefectural Awaji Hospital, Sumoto, Hyōgo
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Kanazawa Medical University Hospital, Nakajima, Ishikawa-ken
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kagawa Medical University Hospital, Kida, Kagawa-ken
  - National Hospital Organization Kagoshima Medical Center, Kagoshima, Kagoshima-ken
  - Kirishima Medical Center, Kirishima, Kagoshima-ken
  - Tokai University Hospital, Isehara, Kanagawa
  - St.Marianna University School Of Medicine Hospital, Kawasaki, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Citizen's General Medical Center attached to Yokohama City University, Yokohama, Kanagawa
  - Kochi Health Sciences Center, Kochi, Kochi
  - Kumamoto Medical University Hospital, Kumamoto, Kumamoto
  - Miyagi Cancer Center, Natori-shi, Miyagi
  - Institute of Development,Aging and Cancer,Tohoku University, Sendai, Miyagi
  - Tohoku University School Of Medicine, Sendai, Miyagi
  - Sendai Medical Center, Sendai, Miyagi
  - Nagano Municipal Hospital, Nagano, Nagano
  - Niigata Prefectural Cancer Center, Niigata, Niigata
  - Kaneda Hospital, Maniwa, Okayama-ken
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Rinku General Medical Center, Izumisano, Osaka
  - Kimen Municipal Hospital, Kimen, Osaka
  - Kitano Hospital, Osaka, Osaka
  - Osaka City University Graduate School of Medicine, Osaka, Osaka
  - Osaka Koseinenkin Hospital, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Sakai Municipal Hospital, Sakai, Osaka
  - Osaka Rosai Hospital, Sakai, Osaka
  - Suita Municipal Hospital Website, Suita, Osaka
  - Yao City Hospital, Yao, Osaka
  - Saga Prefectural Hospital Kouseikan, Saga, Saga-ken
  - Saiseikai Shiga Hospital, Rittō, Shiga
  - Shimane University Faculty of Medicine, Izumo, Shimane
  - Matsue City Hospital, Matsue, Shimane
  - Dokkyo University School of Medecine, Shimotsuga, Tochigi
  - Nippon Medical School, Bunkyo-ku, Tokyo
  - Surugadai Nihon University Hospital, Chiyoda-ku, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Toho University Ohhashi Medical Center, Meguro-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - The Jikei University, Minato-ku, Tokyo
  - International University of Health and Welfare Mita Hospital, Minato-ku, Tokyo
  - Toho University Omori Medical Center, Oota-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Institute of Gastorenterology, Shinjuku-ku, Tokyo
  - Metropolitan Bokutoh Hospital, Sumida-ku, Tokyo
  - Tottori University Faculty of Medicine, Yonago, Tottori
  - Saiseikai Takaoka Hospital, Takaoka, Toyama
  - Kouseiren Takaoka Hospital, Takaoka, Toyama
  - Toyama Prefectural Center Hospital, Toyama, Toyama
  - Yamagata University Faculty Of Medicine, Yamagata, Yamagata

REFERENCES:
- [Derived] Tanabe K, Fujii M, Nishikawa K, Kunisaki C, Tsuji A, Matsuhashi N, Takagane A, Ohno T, Kawase T, Kochi M, Yoshida K, Kakeji Y, Ichikawa W, Chin K, Terashima M, Takeuchi M, Nakajima T. Phase II/III study of second-line chemotherapy comparing irinotecan-alone with S-1 plus irinotecan in advanced gastric cancer refractory to first-line treatment with S-1 (JACCRO GC-05). Ann Oncol. 2015 Sep;26(9):1916-1922. doi: 10.1093/annonc/mdv265. Epub 2015 Jun 24. PMID 26109630